CLINICAL TRIAL: NCT03255200
Title: ReActiv8 Post Market Surveillance Registry for the ReActiv8 Implantable Neurostimulation System for Chronic Low Back Pain
Brief Title: ReActiv8 Post Market Surveillance Registry
Acronym: ReActiv8-C
Status: Completed | Type: Observational
Sponsor: Mainstay Medical (Industry)
Responsible Party: Sponsor
Other Study IDs: 950066
Record Dates: First submitted 2017-08-15; First posted 2017-08-21 (Actual); Results first posted 2024-10-16 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Chronic Low Back Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: ReActiv8 Implantable Stimulation System — Implantable electrical stimulation system.

SUMMARY:
To gather data on the long-term safety of ReActiv8 and identify any residual risks by reporting all Serious Adverse Device Effects as well as performance and health care utilization through two years post-implant.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the Indications for ReActiv8
2. Willing to sign the Informed Consent for the Registry
3. Age ≥ 18 years

Exclusion Criteria:

1. Subjects will be excluded from the Registry if they are contraindicated for ReActiv8.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population for this registry is persons with chronic low back pain who are indicated for ReActiv8.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2023-03-20 (Actual); Study Completion 2023-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schu, MD, Principal Investigator — SANA Klinikum Duisburg
Locations (5):
- Germany (5):
  - Orthopadisches Krankenhaus Schloss Werneck, Werneck, Balthasar-Neumann
  - BG Klinikum Bergmannstrost, Halle
  - Medizinisches Versorgungszentrum Steinburg gGmbH, Itzehoe
  - Katholisches Klinikum Koblenz, Koblenz
  - Klinikum Magdeburg, Magdeburg

RESULTS

PARTICIPANT FLOW:
Groups:
- ReActiv8: All participants implanted with ReActiv8 at baseline.
Period: Overall Study
Arm/Group | ReActiv8
Started | 87
Implanted | 87
Month 3 | 85
Month 6 | 85
Year 1 | 80
Year 2 | 74
Completed | 74
Not Completed | 13

BASELINE CHARACTERISTICS:
Arm/Group | ReActiv8
Number analyzed (Participants) | 87
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (13.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53
  Male | 34
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Germany | 87
Numeric Pain Rating (NRS) Scale [Mean (Standard Deviation); unit: units on a scale] — The Numerical Rating Scale (NRS) is an 11-point scale where 0 means no pain at all and 10 means worst imaginable pain. Patients were asked to rate their average low back pain in the last 24 hours. Lower scores or reduction in score means an improvement or reduction in pain.
  units on a scale | 7.6 (1.2)
Oswestry Disability Index (ODI) [Mean (Standard Deviation); unit: units on a scale] — ODI is a disease specific questionnaire of the disabling effects of back pain and has 10 sections: pain intensity, personal care, lifting, walking, sitting, standing, sleeping, sex life (if applicable), social life, and travelling. Each section has 6 statements correlating to scores of 0 through 5, with the Subject choosing the statement that matches their ability. Scores from 0 to 20% indicate minimal disability; 21-40%, moderate disability; 41-60%, severe disability; 61-80%, crippled; and 81-100%, bedbound or exaggerating. A lower score means an improvement, or reduction in disability.
  units on a scale | 42.4 (15.6)
European Quality of Life - Five Dimensions (EQ-5D) [Mean (Standard Deviation); unit: units on a scale] — The European Quality of Life - Five Dimensions (EQ-5D) is a questionnaire of health-related quality of life consisting of five dimensions (mobility, self-care, usual activities, pain/discomfort, anxiety/depression) each of which can take one of five responses. The responses record five levels of severity (no problems, slight problems, moderate problems, severe problems, extreme problems) within a particular dimension. The EQ-5D Index is scored on a scale from -0.59 to 1.00, with a score of 1.00 indicating full health. A higher score means an improvement in health-related quality of life.
  units on a scale | 0.5 (0.2)
Opioid Use [Count of Participants; unit: Participants] | 26
Pain Duration [Mean (Standard Deviation); unit: years] | 7.7 (7.8)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m 2] | 28.3 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: Low Back Pain - Numeric Pain Rating (NRS) Scale
Description: Change in low back pain Numerical Rating Scale (NRS) compared to Baseline. The NRS is an 11-point scale where 0 means no pain at all and 10 means worst imaginable pain. Patients were asked to rate their average low back pain in the last 24 hours. Lower scores or reduction in score means an improvement or reduction in pain.
Time Frame: 90 days, 180 days, 1 year, 2 years post Activation
Population: Of the 87 patients implanted, 84 completed the Day 3 month, 85 completed the Day 6 month, 79 completed the Year 1 visit, and 74 completed the Year 2 visit. Some patients were withdrawn or lost to follow-up.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | ReActiv8
Number analyzed (Participants) | 87
units on a scale
  Month 3: number analyzed (Participants) | 84
  Month 3 | 4.5 (2.3)
  Month 6: number analyzed (Participants) | 85
  Month 6 | 4.3 (2.6)
  Year 1: number analyzed (Participants) | 79
  Year 1 | 3.8 (2.5)
  Year 2: number analyzed (Participants) | 74
  Year 2 | 3.4 (2.7)

2. Secondary Outcome: Serious Adverse Device Effects
Description: All serious device- or procedure-related adverse events.
Time Frame: Through 2 years post Activation
Measure: Count of Participants; unit: Participants
Arm/Group | ReActiv8
Number analyzed (Participants) | 87
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | ReActiv8
All-Cause Mortality (participants affected / at risk) | 1/87
Serious Adverse Events (participants affected / at risk) | 21/87
Other Adverse Events (participants affected / at risk) | 6/87
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReActiv8 (N=87)
Allergic Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Stomach pain (Gastrointestinal disorders) | 1 (1)
Upper back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myocardial infarction (Cardiac disorders) | 2 (2)
Urinary Tract Infection (Infections and infestations) | 1 (1)
Lung Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Herniated disc (Musculoskeletal and connective tissue disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Radiculopathy (Nervous system disorders) | 1 (1)
Vocal cord paresis (Nervous system disorders) | 1 (1)
Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 (1)
Arterial Bleeding (Vascular disorders) | 1 (1)
Intervertebral Disc Prolapse (Musculoskeletal and connective tissue disorders) | 1 (1)
Gastroenteritis (Gastrointestinal disorders) | 1 (1)
Death; Cause Unknown, Unrelated to Study Treatment (General disorders) | 1 (1)
Shoulder Fracture (Musculoskeletal and connective tissue disorders) | 1 (1)
Overdose (Injury, poisoning and procedural complications) | 1 (1)
Knee pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Hip pain (Musculoskeletal and connective tissue disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ReActiv8 (N=87)
Pain Sacroiliac (Musculoskeletal and connective tissue disorders) | 6 (7)

LIMITATIONS AND CAVEATS:
This study was an open-label registry with no formal statistical hypotheses. The sample size was based on the desire to gain a sufficient amount of representative data with the device in the post-market setting. It provides real-world data on the safety and performance of the device but is not a robust clinical trial, and thus, has the potential for bias.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2020-05-27): https://cdn.clinicaltrials.gov/large-docs/00/NCT03255200/Prot_000.pdf